CLINICAL TRIAL: NCT03370042
Title: Comparative Clinical Evaluation of Semilunar Coronally Positioned Flap Alone and Semilunar Coronally Positioned Flap in Conjunction With Free Gingival Graft for Root Coverage
Brief Title: Single Stage Root Coverage for Gingival Recession With or Without Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kamineni Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, RAGA BINDU, Post Graduate, Kamineni Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBINDU
Record Dates: First submitted 2017-12-02; First posted 2017-12-12 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Gingival Recession
Keywords: aesthetics; root coverage; semilunar coronally positioned flap; free gingival graft; width of keratinised tissue
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semilunar Coronally Positiones Flap + Free Gingival Graft (Active Comparator): semilunar coronally positioned flap with free gingival graft for root coverage
  Interventions: Procedure: semilunar coronally positioned flap with free gingival graft
- Semilunar Coronally Positioned Flap (Sham Comparator): semilunar coronally positioned flap alone without free gingival graft for root coverage
  Interventions: Procedure: semilunar coronally positioned flap alone

INTERVENTIONS:
Procedure: semilunar coronally positioned flap with free gingival graft
  Other Names: combination technique
  Arms: Semilunar Coronally Positiones Flap + Free Gingival Graft
Procedure: semilunar coronally positioned flap alone
  Other Names: pedicle flap
  Arms: Semilunar Coronally Positioned Flap

SUMMARY:
Background and Objective: Gingival recession accounts for apical migration of the gingival margin resulting in exposure of the cementoenamel junction (CEJ) and root surface. It is a matter of concern for both patients and dental professionals, especially when exposure of the root surface is linked to deterioration in esthetic appearance and increase in dentinal hypersensitivity which leads to improvements in various surgical techniques that have been used to correct labial gingival recession defects. The present study thus was aimed to evaluate and compare the results of Semilunar Coronally Positioned Flap alone and Semilunar Coronally Positioned Flap in Conjunction with Free Gingival Graft for treatment of Miller Class I and II gingival recession defects in maxillary anterior teeth.

Materials and Method: A total of 20 bilateral Miller's class I and II gingival recession sites in systemically healthy subjects, 20-45 years of age were recruited for this study. Recession sites were divided and randomly allocated to either of the two groups SCPF+FGG (test group) and SCPF (control group) with 10 sites per group to be treated with semilunar coronally positioned flap with free gingival graft technique for SCPF+FGG group and semilunar coronally positioned flap technique alone for SCPF group. Longitudinal alterations during a follow-up period of 1, 3, 6 and 12 months in terms of Probing depth (PD), Recession width (RW), Recession height (RH), Width of keratinized tissue (WKT) and Clinical attachment level (CAL) were measured for both the groups and the values were statistically analysed.

DETAILED DESCRIPTION:
Gingival recession is a matter of concern for both patients and dental professionals, especially when exposure of the root surface is linked to deterioration in esthetic appearance and increase in dental hypersensitivity which provoked to propose various surgical techniques that have been used to correct labial/buccal gingival recession defects including periodontal plastic surgery. The goal of these surgical procedures is to correct the recession defects and remove or control the etiologic factors that result in mucogingival problems including free gingival autografts,laterally and coronally positioned flap, semilunar flap, guided tissue regeneration(GTR), subepithelial connective tissue graft (SCTG) and combination of procedures.

The selection of surgical technique depends on several factors including the anatomy of the defect site, size of recession defect, presence or absence of keratinized tissue adjacent to the defect, width and height of the interdental soft tissue and depth of the vestibule or the presence of frenula. It also depends on the objective of the treatment outcome which varies in maxilla and in mandible. In maxilla the desired outcome is aesthetics where as in case of mandible it is the mucogingival problems with restoration of normal function. Because of the existing controversies about using different techniques of root coverage and their disadvantages, there are only few documented reports about an esthetic outcome which is important in maxilla that can be gained through increased width of keratinized tissue.

The semilunar coronally positioned flap (SCPF) procedure introduced by Tarnow for treatment of gingival recessions is confined to the maxillary arch with esthetic outcome but no attempt is made to increase the width of keratinized tissueor thickness of gingival tissue. On the other hand, free gingival autograft (FGG) increases the width of keratinized tissue or thickness of gingiva predictably but may result in compromised color match due to lighter color of the graft. Thus simultaneous use of SCPF and FGG was performed to combine both desirable outcomes.

As there are no documented reports about comparative clinical evaluation of SCPF and simultaneous use of SCPF and FGG for covering the exposed root surface in Miller's class I and II gingival recession, an attempt is made to evaluate the results of simultaneous use of SCPF and FGG for covering the exposed root surface and its comparison with SCPF alone in the present study. Thus the aim of the present study is to compare and evaluate the results of using semilunar coronally positioned flap alone for root coverage with a combination technique of semilunar coronally positioned flap along with free gingival graft for root coverage and to assess the results of a combination technique of semilunar coronally positioned flap along with free gingival graft for root coverage. The goal of treatment is to improve aesthetic outcomes with gain in the keratinised tissue levels and clinical attachment level in addition to possible root coverage in maxillary anteriors.

Study Design:

A total of 20 bilateral Miller's class I and II recession sites in maxillary anteriors (incisors or premolars) in systemically healthy subjects, 20-45 years of age, were consecutively recruited from the outpatient department of Periodontology, Kamineni Institiute of Dental sciences, Narketpally, Nalgonda (Dist) who desired treatment for gingival recession in maxillary incisor or premolar area for this study. The study design was approved by the Institutional Ethical Committee, Kamineni Institute of Dental Sciences. The nature and purpose of the study was explained to the patients in their native language and an informed consent was obtained.

Bilateral recession defects in each patient were randomly divided into two groups, SCPF+FGG (test group) who were treated with combined technique of semilunar coronally positioned flap with free gingival graft and SCPF (control group) treated with semilunar coronally positioned flap alone, 10 defects in each group. The defects were randomly selected by coin toss to be treated either with the SCPF + FGG or SCPF alone. Changes in clinical parameters during a follow-up period of 1, 3, 6 and 12 months were recorded using UNC 15 probe along the long axis of the tooth over the mid-root surface expressed in millimetres. An acrylic occlusal stent was used as the fixed reference point to determine the amount of root coverage gained and changes in probing attachment level during the follow up where as WKT assessed using Lugol's iodine.

Initial therapy:

Prior to surgery, all subjects received oral prophylaxis, which included scaling and root planing with ultrasonic instruments (EMS) and Gracey curettes (Hu-Friedy, USA) and crown polishing along with oral hygiene instructions.Only when the patient demonstrated the ability to maintain a good level of oral hygiene was the surgical phase initiated.

SURGICAL PROCEDURE:

Bilateral defects were treated at the same appointment and all the defects were treated by the single person.

Control Group: Semilunar Coronally Positioned Flap (SCPF) Group The operation area was anaesthetized using local anesthesia (2% lignocaine with 1:80000 adrenaline). The exposed root surface was planed to remove altered cementum and flatten it to permit a more intimate adaptation of the flap to the recipient bed. Semilunar incision following the curvature of the free gingival margin is made with No. 15 blade. The incision should curve apically far enough mid-facially to ensure that the apical part of the flap rests on bone after it is brought down to cover the exposed root. The incision should end into the papilla on each end of the tooth,but not all the way to the tip of the papilla. At least 2 mm must be left on either side of the flap (Fig.1-B), since this is the main source of blood supply. Later a sulcular split thickness incision is made.Using microsurgical blades (Lance tip blade 150 and Slit blade 2.8mm), a split thickness dissection is made from the initial incision line coronally. This is connected with an intra-sulcular incision, made mid-facially. The mid-facial tissue is then coronally positioned to the CEJ, or to the height of the adjacent papilla. The tissue is held in place with moist gauze against the tooth for 5 min then sutured with sling sutures using vicryl 5-0 (Fig.1-C). A thin layer of periodontal dressing (Coepack®) was applied over the site.

SCPF+FGG (Test Group): Combined technique of Semilunar coronally positioned flap with Free gingival graft:

After initial semilunar coronally positioned flap similar to SCPF group, the denuded area between the initial incision and the apical margin of the coronally positioned flap is the recipient site for the free gingival graft. A tin foil was placed on the recipient site and a template was prepared. The tin foil template was then placed over the palatal area and an incision was made all round the template to a depth of 2 mm and 1 mm larger than the outline of the tin foil to accommodate graft shrinkage. The harvested graft (Fig.1-D) was placed on to gauze soaked in normal saline solution. The underside of the graft was inspected overhanging tissues. The donor area was then closed with continuous sutures.The graft was adapted to the recipient site and immobilized by holding sutures using 5-0 vicryl suture (Fig.1-E). The graft was firmly held in place using digital pressure for 5 minutes to reduce the dead space, permit fibrin clot formation and prevent bleeding as it may result in a hematoma under the graft and cause subsequent necrosis. Periodontal dressing (Coepack®) was placed at the donor site and over the graft.

Post operative care:

The patients were advised not to brush the treated site for 2 weeks and instead 0.2% chlorhexidine rinse was prescribed for 4 weeks.Antibiotics and analgesics were administered as needed.Then they were examined after 2 weeks to assess healing and removal of sutures. Then after, the patients were instructed to gently brush around the surgical site with an ultra soft toothbrush using roll technique. Routine oral health care was used in other sites. Subjects were enrolled in a follow up program at 1, 3, 6 and 12 months after surgery for the rest of the study. Complete plaque elimination was performed every 3 months.

Stastical Analysis:

Statistical analysis was performed using a commercially available software program (SPSS version 16.0;SPSS, Chicago, IL, USA).Repeated Measure ANOVA was used to investigate whether data were normally distributed or not. The Wilcoxonsigned-ranks test was used for intragroup comparisons and Mann-Whitney U non-parametric test for intergroup comparisons of the clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral Miller Class I and II gingival recessions in maxillary anterior teeth

Exclusion Criteria:

* systemic conditions known to interfere with periodontal healing
* history of addiction or drinking alcohol
* Systemic or local bone diseases
* Pregnancy and lactating females
* using anticoagulant or immune suppressor drugs
* the patients who are unable to maintain oral hygiene
* presence of Type II and V caries and
* smokers

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-14 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-11-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Recession defects
Groups:
- SCPF + FGG: semilunar coronally positioned flap with free gingival graft
  semilunar coronally positioned flap with free gingival graft
- SCPF: semilunar coronally positioned flap alone
  semilunar coronally positioned flap alone
Period: Overall Study
Arm/Group | SCPF + FGG | SCPF
Started | 10; 10 Recession defects | 10; 10 Recession defects
Completed | 10; 10 Recession defects | 10; 10 Recession defects
Not Completed | 0; 0 Recession defects | 0; 0 Recession defects

BASELINE CHARACTERISTICS:
Groups:
- SCPF + FGG: semilunar coronally positioned flap with free gingival graft
- SCPF: semilunar coronally positioned flap alone
- Total: Total of all reporting groups
Arm/Group | SCPF + FGG | SCPF | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Median (Full Range); unit: years] | 32.5 [20 to 45] | 32.5 [20 to 45] | 32.5 [20 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  India | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Recession Height
Description: measured from cemento enamel junction to the most apical part of gingival margin
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SCPF + FGG | SCPF
Number analyzed (Participants) | 10 | 10
mm | 1.0 (1.05) | 0.9 (0.7)

2. Primary Outcome: Width of Keratinized Tissue
Description: measured from most apical part of gingival recession to the mucogingival junction
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SCPF + FGG | SCPF
Number analyzed (Participants) | 10 | 10
mm | 4.7 (1.07) | 3.6 (0.84)

3. Secondary Outcome: Clinical Attachment Level
Description: combined probing depth and recession height
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SCPF + FGG | SCPF
Number analyzed (Participants) | 10 | 10
mm | 2.4 (0.9) | 2.3 (1.05)

4. Secondary Outcome: Probing Depth
Description: gingival margin to the base of the sulcus
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- SCPF + FGG: semilunar coronally positioned flap with free gingival graft for root coverage
- SCPF: semilunar coronally positioned flap alone without free gingival graft for root coverage
Arm/Group | SCPF + FGG | SCPF
Number analyzed (Participants) | 10 | 10
mm | 1.3 (0.4) | 1.3 (0.4)

5. Secondary Outcome: Recession Width
Description: mesial gingival margin to distal gingival margin at cemento enamel junction
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SCPF + FGG | SCPF
Number analyzed (Participants) | 10 | 10
mm | 1.3 (1.3) | 1.4 (1.07)

ADVERSE EVENTS:
Description: Adverse effects not monitored or assessed
Arm/Group | SCPF + FGG | SCPF
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The stabilisation of the donor graft with sutures over the recipient bed as it requires exceedingly small section of donor tissue. FGG placed apical to the flap may undergo shrinkage affecting the root coverage on long term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2014-12-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT03370042/ICF_000.pdf